CLINICAL TRIAL: NCT05056142
Title: Epidural Versus Low-dose Spinal for Analgesia of Late First Stage of Labor: A Randomized Clinical Trial
Brief Title: Epidural Versus Low-dose Spinal for Analgesia of Late First Stage of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amin Mohammed Alansary Amin Ahmed Helwa, Associate Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: FMASU R 155/2021
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Anesthesia, Epidural

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural Anesthesia (Active Comparator): Patients will receive epidural analgesia with 15 ml isobaric bupivacaine 0.125% plus fentanyl 2 μg/mL
  Interventions: Procedure: Epidural Anesthesia
- Spinal Anesthesia (Active Comparator): Patients will receive Spinal analgesia with 5 mg bupivacaine and 25 μg of fentanyl in a 2 ml volume.
  Interventions: Procedure: Spinal Analgesia

INTERVENTIONS:
Procedure: Epidural Anesthesia — Patients will receive epidural analgesia with 15 ml isobaric bupivacaine 0.125% plus fentanyl 2 μg/mL.
  Arms: Epidural Anesthesia
Procedure: Spinal Analgesia — Patients will receive Spinal analgesia with 5 mg bupivacaine and 25 μg of fentanyl in a 2 ml volume.
  Arms: Spinal Anesthesia

SUMMARY:
The aim of this study is to compare the effect of epidural analgesia versus low-dose spinal analgesia in parturient in the late first stage of labor regarding time needed to perform the block, duration of the intra- and postoperative analgesia and incidence of procedure related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Parturient with normal vaginal delivery in late first stage of labor (cervical dilatation ≥ 6 cm by examination)
* Aged 18-40 years old
* Single, term pregnant with normal fetal heart rate
* Request neuroaxial analgesia

Exclusion Criteria:

* Parturient who refuses to participate,
* American Society of Anesthesiologists (ASA) physical status >II,
* Body mass index more than 35 kg/m2
* Severe pre-eclampsia or eclampsia
* Uncontrolled thyrotoxicosis
* Cardiovascular troubles (e.g. stenotic valvular heart disease or cardiomyopathy)
* Increased intracranial tension due to a space-occupying lesion
* Any contraindication to regional anesthesia such as local skin or soft tissue infection, coagulopathy or receiving anticoagulant therapy, thrombocytopenic, uncorrected hypovolemia, preexisting neurologic deficits, spinal deformity or previous spine surgery.
* Hypersensitivity to the study drugs
* Parturient who scheduled for emergency cesarean section due to fetal distress, antepartum hemorrhage, multiple gestation or fetal malpresentation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
The time to perform the block | Intraoperative
  The time from the preparation of the block until the full injection of anesthetic drugs,

SECONDARY OUTCOMES:
Mean arterial blood pressure (MAP) | Intraoperative
  MAP will be recorded at baseline; 5 minutes prior to the neuroaxial block, and at 5 minutes, 10 minutes, 15 minutes, and 20 minutes after the injection of the local anesthetic and then every 15 minutes till the end of third stage of labor
Heart rate (HR) | Intraoperative
  HR will be recorded at baseline; 5 minutes prior to the neuroaxial block, and at 5 minutes, 10 minutes, 15 minutes, and 20 minutes after the injection of the local anesthetic and then every 15 minutes till the end of third stage of labor
Number of participnts with Postoperative nausea and vomiting (PONV) | First 24 hours postoperatively
  PONV will be recorded and categorized as 'no PONV, mild PONV, moderate PONV, and severe PONV'

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided